CLINICAL TRIAL: NCT03215017
Title: A Randomized Controlled Study of the Effect of Treatment of Low Anterior Resection Syndrome (LARS) After Rectal Cancer Surgery
Brief Title: Effect of Treatment of Low Anterior Resection Syndrome After Rectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mirna Abraham-Nordling (Other)
Responsible Party: Sponsor-Investigator, Mirna Abraham-Nordling, MD. PhD. Associate Professor of Surgery, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/551-31
Record Dates: First submitted 2017-07-01; First posted 2017-07-12 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome | interventions — Dosage Forms; Sorbitol; Karaya Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transanal irrigation (Experimental): Manual transanal irrigation to control bowel function.
  Interventions: Device: Transanal irrigation
- Medication (Active Comparator): Medication to control bowel function.
  Interventions: Drug: Medication

INTERVENTIONS:
Device: Transanal irrigation — Effect of Transanal irrigation (TAI) using Peristeen® anal irrigation system - Coloplast
  Other Names: Peristeen® anal irrigation system - Coloplast
  Arms: Transanal irrigation
Drug: Medication — Medication to help control of the bowel movement (One or a combination of Loperamide, Sorbitol, Sterculia gum)
  Other Names: One or a combination of Loperamide, Sorbitol, Sterculia gum
  Arms: Medication

SUMMARY:
A randomized controlled trial (RCT) in patients who underwent sphincter preserving surgery due to rectal cancer. The study will analyze the effect of Transanal irrigation (TAI) and medication that can help control of the bowel movement in patients with low anterior resection syndrome.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) in patients who underwent sphincter preserving surgery due to rectal cancer.

The study will analyze the effect of Transanal irrigation (TAI) and medication that can help control of the bowel movement in patients with low anterior resection syndrome.

An interim analysis will be made after 40 included patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have undergone surgery for rectal cancer (sphincter saving surgery, low anterior resection)
* Adult ≥ 18 years old
* Have scoring major LARS (according to the Low anterior resection syndrome score)

Exclusion Criteria:

* stoma
* recurrent disease
* Another colorectal surgery
* Inflammatory bowel disease (IBD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Bowel function | 1 year
  Cleveland incontinence questionnaire
Bowel function, Low anterior resection syndrome (LARS) | 1 year
  Assessed using LARS questionnaire (score 0-42, a high score indicates poor bowel function)

SECONDARY OUTCOMES:
Quality of Life (QoL) | 1 year
  Assessed using EORTC Quality of life questionnaire (QLQ)-C30

CONTACTS AND LOCATIONS:
Overall Officials: Mirna Abraham-Nordling, MD.PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Danderyd Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Stockholm South General Hospital, Stockholm

REFERENCES:
- [Background] Pieniowski EHA, Bergstrom CM, Nordenvall CAM, Westberg KS, Johar AM, Tumlin Ekelund SF, Larsson KR, Pekkari KJ, Jansson Palmer GC, Lagergren P, Abraham-Nordling M. A Randomized Controlled Clinical Trial of Transanal Irrigation Versus Conservative Treatment in Patients With Low Anterior Resection Syndrome After Rectal Cancer Surgery. Ann Surg. 2023 Jan 1;277(1):30-37. doi: 10.1097/SLA.0000000000005482. Epub 2022 Jul 7. PMID 35797618